CLINICAL TRIAL: NCT06988917
Title: Rehabilitation Efficacy of Low-Load Blood Flow Restriction Training for Lateral Patellar Compression Syndrome
Acronym: LL-BFRT
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024150
Record Dates: First submitted 2025-04-29; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-03

CONDITIONS: Lateral Patellar Compression Syndrome
Keywords: Lateral Patellar Compression Syndrome; patellofemoral joint; LL-BFRT

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — Age, Body Mass Index (BMI), Gender, Site of Injury, and Combined Meniscal Injury
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The experimental group (LL-BFRT group): The experimental group (LL-BFRT group) received exercise intervention treatment for 4 weeks, training three times a week, each time lasting for 1 hour. Compared with the control group (conventional rehabilitation group), the movements and intensities of the two groups remained consistent during the exercise intervention. Only the experimental group wore a flow-limiting pressure band for exercise during the intervention. The blood flow limiting pressure band used in this study mainly consists of a 109*10cm leg pressure band, a barometric display dial with a pressure range of 0-300mmHg, and a pressure pump. In the experiment, we fixed the blood flow restriction pressure band in the area for measuring the circumference and adjusted the blood flow restriction pressure according to the thigh circumference of the subjects to maintain it within the range of 40%-60% arterial occlusion pressure. The way to limit blood flow is intermittent inflation.
  Interventions: Behavioral: the regular rehabilitation program; Device: The blood flow limiting pressure band
- The control group (conventional rehabilitation group): The control group (conventional rehabilitation group) received exercise intervention treatment for 4 weeks, with training three times a week, each lasting for 1 hour. The specific intervention contents are: Each training session consists of a 10-minute warm-up (including power cycling, full-body stretching, etc.) At the same time, use the foam axis to relax the lateral oblique femoris and iliotibial band to relieve the pressure on the lateral side of the patella), 40 minutes of formal training (including wall squats with a ball, straight leg raising resistance training, terminal resistance knee extension training, bench kick ball clamping training, and balance training), and 10 minutes of relaxation (using a foam roller, foam axis and other combined techniques to relax the muscles Especially for the lower limb muscles such as the lateral femoris, iliotibial band, and tibialis anterior muscle.
  Interventions: Behavioral: the regular rehabilitation program

INTERVENTIONS:
Behavioral: the regular rehabilitation program — Each training session consists of a 10-minute warm-up (including power cycling, full-body stretching, etc.) At the same time, use the foam axis to relax the lateral oblique femoris and iliotibial band to relieve the pressure on the lateral side of the patella), 40 minutes of formal training (including wall squats with a ball, straight leg raising resistance training, terminal resistance knee extension training, bench kick ball clamping training, and balance training), and 10 minutes of relaxation (using a foam roller, foam axis and other combined techniques to relax the muscles Especially for the lower limb muscles such as the lateral femoris, iliotibial band, and tibialis anterior muscle.
Device: The blood flow limiting pressure band — The experimental group (LL-BFRT group) wore a flow-limiting pressure band for exercise during routine rehabilitation training. The blood flow limiting pressure band used in this study mainly consists of a 109*10cm leg pressure band, a barometric display dial with a pressure range of 0-300mmHg, and a pressure pump. In the experiment, we fixed the blood flow restriction pressure band in the area for measuring the circumference and adjusted the blood flow restriction pressure according to the thigh circumference of the subjects to maintain it within the range of 40%-60% arterial occlusion pressure. The way to limit blood flow is intermittent inflation, that is, during the intervals of muscle strength training, the cuff deflation operation is carried out simultaneously.
  Groups: The experimental group (LL-BFRT group)

SUMMARY:
The purpose of this study is to understand the effect of low-load blood flow restriction training on the rehabilitation effect of patients after lateral patellar compression syndrome surgery, and to observe the differences between low-load blood flow restriction training combined with conventional rehabilitation training and conventional rehabilitation training. The main question it aims to answer is:

Can low-load blood flow restriction training improve the rehabilitation effect of patients after surgery for lateral patellar hypertension syndrome? Researchers compared conventional rehabilitation training with conventional rehabilitation training combined with low-load blood-limiting training to explore the effect of blood-limiting training combined with conventional rehabilitation training on the lower extremity function of patients after lateral patellar compression syndrome surgery, providing experimental and theoretical basis for formulating rehabilitation training programs.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 30-60 years with a Visual Analog Scale (VAS) score ≥3;
2. Diagnosed with lateral patellar compression syndrome confirmed by MRI and clinical evaluation, having undergone arthroscopic lateral retinacular release surgery;
3. Presenting postoperative reduction in thigh circumference on the affected side, accompanied by quadriceps muscle atrophy and decreased muscle strength;
4. Minimum postoperative duration of ≥2 weeks, with signed informed consent and demonstrated ability to comply with the study protocol.

Exclusion Criteria:

1. Patients with concomitant fractures or other ligament injuries (including those with prior ACL reconstruction);
2. Individuals presenting with severe osteoarthritis or rheumatoid arthritis;
3. Those with medical histories of deep vein thrombosis, coagulation disorders, vascular diseases, or diabetes mellitus;
4. Subjects with active infections, malignancies, current pregnancy, or psychiatric disorders.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with lateral patellar compression syndrome after lateral retinacular release
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Lysholm score | 0-4week
VAS score | 0-4week
Peak torque of knee extension | 0-4week
Quadriceps thickness | 0-4week

SECONDARY OUTCOMES:
Thigh circumference | 0-4week
Range of motion of the knee joint | 0-4week

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Yang, Principal Investigator
Locations (1):
- Peking University Third Hospital of Chongli, Chongli, Hebei, China